CLINICAL TRIAL: NCT02228226
Title: Follow-up Study After Arthroscopic Bankart Repair Using MG-1 for Dislocation of Shoulder
Brief Title: Follow-up Study After Bankart Repair Using MG-1
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson K.K. Medical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: JJKK-MIT-002
Record Dates: First submitted 2014-08-20; First posted 2014-08-28 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Shoulder Dislocation
Keywords: Arthroscopic Bankart repair; Bone hole; Ossification; Suture anchor; Shoulder dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MG-1treated group: MG-1treated group: Patients those who underwent arthroscopic Bankart repair for glenohumeral instability using MG-1

SUMMARY:
Long term follow-up of patients those who underwent arthroscopic Bankart repair using MG-1 for dislocation of shoulder to evaluate anchor bone hole condition and ossification.

ELIGIBILITY:
Inclusion Criteria:

* Patient who was enrolled to the clinical trial of MG-1 at Funabashi Orthopaedic Hospital and who don't withdraw the consent
* Patient who understand the contents of the study and from whom a written consent can be obtained

Exclusion Criteria:

* Patient with dementia
* Patient who cannot undergo CT examination
* Patient who underwent further surgery to ipsilateral shoulder joint after the clinical trial
* Patient who is pregnant or lactating
* Patient judged to be inappropriate for the study by the (sub)investigator

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients those who underwent arthroscopic Bankart repair for glenohumeral instability using MG-1
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Bone Hole Condition | over 24 months after surgery
  To evaluate Bone Hole Condition with score based on CT images. CT images are evaluated and scored by three evaluators who are MDs and independent of this study director.
  Definitions of the score are described as below.
  * Type 1: Opened or enlarged
  * Type 2: Slightly closed (<50%)
  * Type 3: Almost closed (>=50%)
  * Type 4: Completely closed
Ossification | over 24 months after surgery
  To evaluate Ossification with score based on CT images. CT images are evaluated and scored by three evaluators who are MDs and independent of this study director.
  Definitions of the score are described as below.
  * Type 1: Little or no ossification
  * Type 2: Ossification fills some of the anchor site that is discontinuous or with a wide lucent rim
  * Type 3: Ossification fills most of the anchor site with a thin lucent rim. This area's density is consistent with cancellous bone
  * Type 4: Ossification fills the anchor site completely with an indistinct border between the anchor site and the adjacent cancellous bone

SECONDARY OUTCOMES:
Clinical Function Evaluation | over 24 months after surgery
  To evaluate the Japan Shoulder Society Shoulder Instability Score (JSS-SIS) and Rowe Score at 12 weeks after surgery
  JSS-SIS Score (subscales are summed, higher values represent a better outcome):
  * Pain (0 to 20)
  * Function (0 to 20)
  * Range of Motion (0 to 20)
  * Evaluation of X-ray findings (0 to 10)
  * Stability (0 to 30)
  Rowe Score (subscales are summed, higher values represent a better outcome):
  * Stability (0 to 50)
  * Motion (0 to 20)
  * Function (0 to 30)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroyuki Sugaya, MD, Ph. D, Principal Investigator — Funabashi Orthopaedic Hospital
Locations (1):
- Funabashi Orthopaedic Hospital, Funabashi, Chiba, Japan